CLINICAL TRIAL: NCT02529280
Title: Choices: Increasing Access of Latinas Into Breast Cancer Clinical Trials
Brief Title: Choices for Latinas and Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Amelie Ramirez, Chair, ad interim, and Professor, Department of Epidemiology and Biostatistics, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20090165H
Record Dates: First submitted 2015-08-11; First posted 2015-08-20 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Latinas; Breast Cancer; Clinical Trials; Participation
MeSH Terms: conditions — Breast Neoplasms | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive three components: 1) a culturally sensitive, individually tailored, 30-minute computer-based BCCT video; 2) a bilingual, low-literacy booklet aimed at encouraging patients to communicate with family and friends and 3) assistance from a patient navigator.
  Interventions: Behavioral: Intervention
- Usual Care (No Intervention): The usual care control group will receive the usual care breast cancer clinical trial information materials offered by the CTRC to their eligible patients.

INTERVENTIONS:
Behavioral: Intervention — Intervention includes 1) a 30-minute computer-based video (in English/Spanish), featuring instructional screens, graphics and animation to help participants understand the concepts presented. It will feature breast cancer patients who have participated in CTs, patients talking to their doctor or nurse and a bilingual narrator to guide participants. Video content will address common barriers and concerns regarding clinical trials, as well as the informed consent process, and how clinical trials are monitored and reviewed; 2) a bilingual easy to understand booklet with tailored information on clinical trials. The booklet will include many of the elements and messages featured in the video program; and 3) assistance from a trained, bilingual, bicultural, nurse navigator.
  Arms: Intervention

SUMMARY:
"Increasing Access of Latinas into Breast Cancer Clinical Trials" aims to develop and pilot test a multi-communications approach - using a culturally relevant computer video, a tailored booklet and a patient navigator (PN) - to empower Latinas to make informed decisions about breast cancer clinical trials (BCCTs). Latinos represent 15% of the U.S. population but only 5.6% of participants in National Cancer Institute (NCI) treatment clinical trials, resulting in disparities in cancer outcomes and jeopardizing the generalizability of trial findings. In response, this study will develop and evaluate communication and health-system-change strategies to facilitate Latinas' access to BCCTs at the Cancer Therapy and Research Center at The University of Texas Health Science Center at San Antonio (CTRC-UTHSCSA). The CTRC-UTHSCSA, an NCI-designated Cancer Center located in South Texas, serves a culturally and ethnically diverse population that historically has low participation in clinical trials, especially among those with breast cancer, the No. 1 cancer killer of Latinas.

DETAILED DESCRIPTION:
This study features a cohort design with random assignment of 112 Latina breast cancer patients from the CTRC to an intervention (56) or usual care control group (56). The intervention group will receive three components: 1) a culturally sensitive and individually tailored, 30-minute computer-based BCCT educational video; 2) a bilingual, low literacy booklet that encourages patients to communicate with family and friends; and 3) support from a patient navigator. The usual care control group will receive usual care breast cancer clinical trial information materials offered by the CTRC to its eligible patients. The intervention is based in two proven theories - Stages of Change and Social Cognitive Theory - and will feature basic components of individual empowerment, including knowledge, attitudes, skills and self-efficacy beliefs and expectations.

The study has three main phases: Phase 1: Formative Research; Phase 2: Intervention; and Phase 3: Evaluation.

Purpose:

To empower Latinas to make informed decisions about breast cancer clinical trials (BCCTs) by enhancing their knowledge, attitudes, skills and self-efficacy required to support discussion of CT as a treatment option with doctors and family members.

Specific Objectives:

1. Increase patient education and awareness, positive attitudes and self-efficacy to enhance their decision-making skills to participate in BCCTs.
2. Provide decisional support to make an informed decision regarding participation in BCCTs by encouraging discussion of BCCTs as a treatment option with medical team, family and friends.
3. Test the efficacy of a multi-communication intervention to assist Latina breast cancer patients in their decision making process regarding participation in BCCTs.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking Latinas diagnosed with breast cancer who: attend the CTRC breast clinic and/or other CTRC clinics, have not had their initial doctor consultation to discuss treatment options, have not participated in a clinical trial before, and are eligible to participate in one of the Phase III, Phase IV or selective Phase II breast cancer clinical trials (BCCT) open at the CTRC at the time of diagnosis.

Exclusion Criteria:

* Non-Hispanic women
* Children
* Men

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Attitudes towards clinical trials | Baseline and post intervention survey within 3 months from baseline
  Eight-item scale measuring attitudes towards clinical trials (staging questions)
Self-efficacy | Baseline and post intervention survey within 3 months from baseline
  14-item scale measuring self-efficacy regarding seeking information about clinical trials, communication with doctors, family members and friends, confidence in the system, decision making and expectations if enrolled in a clinical trial.
Enrollment in a Clinical Trial | within 6 months from baseline
  Participants' medical records will be reviewed to determine enrollment in a CT

CONTACTS AND LOCATIONS:
Overall Officials: Amelie G. Ramirez, DrPH, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Cancer Therapy and Research Center - CTRC, San Antonio, Texas, United States

REFERENCES:
- [Background] Chalela P, Muñoz E, Gallion JK, Karnad A, Ramirez AG. Empowering Latina breast cancer patients to make informed decisions about clinical trials: A multicommunication approach. Cancer Epidemiol Biomarkers Prev 24(10 Suppl), 2015 [abstract]